CLINICAL TRIAL: NCT03820245
Title: Short-term Annatto Carotenoids Supplementation Effect on LDL Susceptibility to Ex-vivo Oxidation and Oxidative Stress Biomarkers in Healthy Individuals
Brief Title: Effect of Short-term Annatto Carotenoids Supplementation on Oxidative Stress Status in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Lisiane Conte, Master's degree student, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 68801917.0.0000.5346
Record Dates: First submitted 2018-10-19; First posted 2019-01-29 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Oxidative Stress; Atherosclerosis
Keywords: Carotenoid; LDL oxidation; Cardiovascular disease; Antioxidant
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — bixin; norbixin; Lycopene

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bixin (Experimental): Consumption of 0.05 mg bixin/kg b.w. through capsules (once a day) by 7 days in the morning.
  Interventions: Dietary Supplement: Bixin
- Norbixin (Experimental): Consumption of 0.05 mg norbixin/kg b.w. through capsules (once a day) by 7 days in the morning.
  Interventions: Dietary Supplement: Norbixin
- Lycopene (Active Comparator): Consumption of 0.05 mg lycopene/kg b.w. through capsules (once a day) by 7 days in the morning.
  Interventions: Dietary Supplement: Lycopene
- Placebo (Placebo Comparator): Consumption of 0.05 mg placebo/kg b.w. through capsules (once a day) by 7 days in the morning.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bixin — Volunteers consumed bixin capsules during 1 week , maintaining their usal lifestyle (avoiding excessive/unusual of fat and carotenoid-containing food, alcohol)
  Arms: Bixin
Dietary Supplement: Norbixin — Volunteers consumed norbixin capsules during 1 week , maintaining their usal lifestyle (avoiding excessive/unusual of fat and carotenoid-containing food, alcohol)
  Arms: Norbixin
Dietary Supplement: Lycopene — Volunteers consumed lycopene capsules during 1 week , maintaining their usal lifestyle (avoiding excessive/unusual of fat and carotenoid-containing food, alcohol)
  Arms: Lycopene
Dietary Supplement: Placebo — Volunteers consumed placebo capsules during 1 week , maintaining their usal lifestyle (avoiding excessive/unusual of fat and carotenoid-containing food, alcohol)
  Arms: Placebo

SUMMARY:
Low-density lipoprotein (LDL) oxidation has a pivotal role in atherosclerosis development. There is a relationship between carotenoids serum concentration and cardiovascular (CV) benefits, mainly in oxidized LDL (oxLDL) reduction. Despite cardio protective effects of annatto carotenoids, bixin and norbixin, in vitro and in animal studies, its short or long-term supplementation effect on humans are not know. Objective: To analyse CV benefits of annatto carotenoids short-term supplementation in healthy individuals, comparing to lycopene effect. Methods: 16 healthy volunteers (8 men and 8 women) consumed 0.05 mg/kg b.w. of each treatment (bixin, norbixin, lycopene or placebo) through capsules, during 7 days. It was analysed the susceptibility of LDL to Cu2+-induced oxidation, biochemical parameters and oxidative stress biomarkers at the beginning and end of each treatment.

DETAILED DESCRIPTION:
Graduate and post-graduate students were recruited in Federal University of Santa Maria to study participation. First, the health status of volunteers was analysed by questioner application (to evaluate lifestyle, family history, individual characteristics), anthropometric (height, weight, waist circumference) and biochemical parameters (glucose, lipid profile, transaminases, urea, creatinine) measurements. According to inclusion criteria, 18 volunteers were able to study participation, but just 16 people remained until the end of the study.

Each treatment was composed by 7 capsules (containing 0.05 mg carotenoid or placebo/kg b.w.) which should be consumed once a day (preferably in the morning), during 7 days. It was conducted a randomized, double blind, placebo-controlled crossover clinical trial, where 16 participants received 4 proposed treatments (bixin, norbixin, lycopene and placebo) in different periods. To plasma, serum and red blood cells (RBC) obtainment, 2 fasting blood collections were made, in the beginning (Day 0) and the end (Day 7) of each treatment. These samples were used for evaluating the ex vivo oxidation of LDL induced by copper sulphate and biochemical and oxidative biomarkers measurements.

ELIGIBILITY:
Inclusion Criteria:

* Normal levels of glucose, lipid profile, transaminases, urea and creatine
* Normal blood pressure, weight and body mass index (BMI)

Exclusion Criteria:

* Chronic diseases (diabetes, dyslipiademia, hypertension cancer, etc.)
* Drug, alcohol and cigarette consumption/addiction
* Medication, vitamins or suplements consumption (except oral contraceptive used by women)
* Recent inflammatory/infectious diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of LDL lipid moiety susceptibility to copper induced oxidation - oxidation rate | Day 0 and Day 7
  Change (Day 7 - Day 0) of oxidation rate of conjugated dienes formed after copper sulphate addition to LDL particles
Evaluation of LDL protein moiety susceptibility to copper induced oxidation | Day 0 and Day 7
  Evaluate the change (Day 7 - Day 0) of loss of tryptophan fluorescence after oxidation induced by copper
Evaluation of LDL lipid moiety susceptibility to copper induced oxidation - lag phase | Day 0 and Day 7
  Change (Day 7 - Day 0) of lag phase time of conjugated dienes formed after copper sulphate addition to LDL particles

SECONDARY OUTCOMES:
Evaluation of protein oxidation | Day 0 and Day 7
  Change at advanced oxidation protein products levels in plasma
Evaluation of lipid oxidation | Day 0 and Day 7
  Change at malondialdehyde levels in plasma and red blood cells
Evaluation of nitric oxide metabolites | Day 0 and Day 7
  Change at nitric oxide metabolites levels in serum
Evaluation of plasma antioxidant capacity | Day 0 and Day 7
  Change at oxygen radical absorbance capacity in plasma
Evaluation of enzymatic antioxidant defences | Day 0 and Day 7
  Change at antioxidant enzymes activities in red blood cells
Evaluation of gluthatione cycle | Day 0 and Day 7
  Change at reduced glutathione/oxidized glutathione ratio in red blood cells
Evaluation of red blood cell osmotic fragility | Day 7
  Change of red blood cell osmotic fragility after ex vivo exposure to membrane damage inducers
Evaluation of carotenoids levels | Day 0 and Day 7
  Change at carotenoids levels in plasma and red blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Emanuelli, Doctor, Study Director — Universidade Federal de Santa Maria
Locations (1):
- Universidade Federal de Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared after article publication.